CLINICAL TRIAL: NCT04721158
Title: IMPlementation of Continuous Glucose Monitoring in Children With Type 2 Diabetes
Brief Title: CGM Use in Children With Type 2 Diabetes
Acronym: IMPaCT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00255470-2
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes; Hyperglycemia Due to Type 2 Diabetes Mellitus
Keywords: continuous glucose monitoring (CGM); Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CGM Arm (Other): Children with type 2 diabetes will wear a continuous glucose monitor for 10 days.
  Interventions: Device: Continuous glucose monitor

INTERVENTIONS:
Device: Continuous glucose monitor — Eligible patients will have a Dexcom G6 Continuous Glucose Monitor placed for 10 days.
  Other Names: Dexcom G6 CGM

SUMMARY:
The purpose of this prospective study is to determine if trial use of a Dexcom G6 CGM system for a 10 day wear period in pediatric Type 2 diabetes patients improves short term time in range glucose control and 3-6 month glycemic control.

DETAILED DESCRIPTION:
The purpose of this prospective study is to determine if trial use of a Dexcom G6 CGM system for 10 days has an impact on short and long term glycemic control and behavior in youth onset Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, diabetes duration >3 months

Exclusion Criteria:

* Prior use of CGM

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Risa M Wolf, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Pediatric Diabetes Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phu A, Lin T, Manfredo JA, Brown EA, Wolf RM. Similar Perceptions on Continuous Glucose Monitor Use amongst Youth with Type 1 and Type 2 Diabetes. Pediatr Diabetes. 2023 Jun 19;2023:1979635. doi: 10.1155/2023/1979635. eCollection 2023. PMID 40303266

RESULTS

PARTICIPANT FLOW:
Groups:
- CGM Sample Given: Youth with T2D > 3 months, on insulin, with no prior CGM use were enrolled
Period: Overall Study
Arm/Group | CGM Sample Given
Started | 41
Completed | 36
Not Completed | 5
Not completed — Lost to Follow-up | 4
Not completed — Device did not connect | 1

BASELINE CHARACTERISTICS:
Arm/Group | CGM Arm
Number analyzed (Participants) | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16.2 [15 to 17.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 34
  White | 4
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 41
HbA1c [Median (Inter-Quartile Range); unit: Percentage of glycosylated hemoglobin] | 10.3 [7.3 to 12.5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Range Glucose Control
Description: The percentage of total time that the patient uses the continuous glucose monitor (CGM) where the blood glucose falls between 70 and 180 mg/dL
Time Frame: 5 days, 10 days
Population: Participants with CGM use at both 5-days and 10-days
Measure: Mean (Standard Deviation); unit: percentage of time in target range
Arm/Group | CGM Sample Given
Number analyzed (Participants) | 18
percentage of time in target range
  5 days | 49.2 (38)
  10 days | 50.7 (39)

2. Primary Outcome: Hemoglobin A1c
Description: HbA1c at baseline and 3-6 month follow-up.
Time Frame: Baseline, 3 - 6 months
Population: Participants with A1c available at baseline and 3-6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin A1
Arm/Group | CGM Sample Given
Number analyzed (Participants) | 30
percentage of glycosylated hemoglobin A1
  Baseline | 10.2 (2.8)
  3-6 months | 10.3 (3.2)

3. Primary Outcome: More Frequent Insulin Administration
Description: Response to "Did you take your insulin more often than before?"
Time Frame: 10 days from CGM placement
Population: Participants with 10 day follow up surveys
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Arm
Number analyzed (Participants) | 24
Participants
  Yes | 14
  No | 8
  Sometimes | 2

4. Primary Outcome: More Frequent Glycemic Control Monitoring
Description: Response to "Do you look at or check your blood sugar more often than before?"
Time Frame: 10 days
Population: Participants who responded to the survey conducted at 10 day follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | CGM Arm
Number analyzed (Participants) | 24
Participants
  Yes | 23
  No | 0
  Sometimes | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CGM Arm
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 2/41
Other Adverse Events (participants affected / at risk) | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGM Arm (N=41)
DKA admission (Endocrine disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The limitations of this study include the small study size with a limited number of participants completing both 10-day trial period and 3/6-month follow up visits. There were a large number of patients who had device connectivity and adhesive issues. Many participants were lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT04721158/Prot_SAP_000.pdf